CLINICAL TRIAL: NCT03345251
Title: Physical Endometrial Manipulation and Its Effect on Success Rate in Patients With Previous ICSI Failure
Brief Title: Physical Endometrial Manipulation and Its Effect on ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Mahmoud Alalfy, Aljazeera Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Algazeerah
Record Dates: First submitted 2017-10-25; First posted 2017-11-17 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Infertility
Keywords: ICSI - physical - Manipulation - scratching
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: 640 were enrolled but 608 were analyzed
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manipulation of endometrium (Experimental): The arm is physical manipulation to the endometrium prior to ICSI By one of these interventions )Hydrotubation , Sonohysterography or endometrial scratching
  Interventions: Device: Hydrotubation
- no manipulation to endometrium in ICSI (Placebo Comparator): This is the control group , with no manipulation to endometrium prior to ICSI No intervention to this group
  Interventions: Device: Hydrotubation

INTERVENTIONS:
Device: Hydrotubation
  Other Names: Sonohysterography; Endometrial scratching

SUMMARY:
Unexplained infertility is clinically diagnosed when there are no apparent or clear factors causing infertility on regular infertility assessment tools . Failure of implantation is a possible factor causing unexplained infertility . Implantation is the main rate limiting step in IVF outcome. Implantation is described at cellular and molecular level by adhesion or fixation of good quality embryo to receptive endometrium within a critical period of time which is called the window of implantation .

DETAILED DESCRIPTION:
Testing the effect of Physical manipulation of the endometrium on the quality of the endometrium prior to ICSI cycle and if it increases the success rate

ELIGIBILITY:
Inclusion Criteria:

* Infertile female age 20-35 years
* Previous Failed one ICSI trial
* normal basal hormonal profile [FSH, LH] 3-10 mIU/ml and 1.8-8.5 mIU/ml respectively, --normal endometrial cavity
* patent tubes
* normal Husband semen analysis

Exclusion Criteria:

* Ovarian factor of infertility
* Tubal factor of infertility
* Endometrial factor of infertility
* Male factor of infertility

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 640 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-12-25 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
The number of participants who achieved clinical pregnancy | 6 weeks after embryo transfer
  Describes how many participant will continue pregnancy after positive pregnancy test

SECONDARY OUTCOMES:
The number of participants who achieved ongoing pregnancy and live birth | 9 months after embryo transfer
  Describes who many participant will continue pregnancy till he had birth and a live birth

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, master, Study Chair — Algazeerah hospital -Location (Giza -Egypt )
Locations (1):
- Algazeerah, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No